CLINICAL TRIAL: NCT03164486
Title: First-in-Human Positron Emission Tomography Study Using the 18F-αvβ6-Binding-Peptide
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Julie L. Sutcliffe, Ph.D (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Julie L. Sutcliffe, Ph.D, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970652; NCI-2017-00411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCHO028 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma; Lung Carcinoma; Metastatic Malignant Neoplasm in the Breast; Metastatic Malignant Neoplasm in the Colon; Metastatic Malignant Neoplasm in the Lung; Metastatic Malignant Neoplasm in the Rectum; Pancreatic Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-αvβ6-BP (Experimental): Patients receive 18F-alphavbeta6-BP IV and then undergo 4 PET scans over 30 minutes each at 30, 60, 120, and 180 minutes post-injection.
  Interventions: Drug: 18F-αvβ6-BP

INTERVENTIONS:
Drug: 18F-αvβ6-BP — Subjects will be injected once with up to 10 mCi of 18F-αvβ6-BP as a rapid intravenous bolus (within 30 seconds).
  Other Names: Image Enhancement Agent

SUMMARY:
This clinical trial studies the side effects of 18F-alphavbeta6-binding-peptide and how well it works in imaging patients with primary or cancer that has spread to the breast, colorectal, lung, or pancreatic. Radiotracers, such as 18F-alphavbeta6-binding-peptide, may improve the ability to locate cancer in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, biodistribution and dosimetric properties of 18F-alphavbeta6-binding peptide (BP) in normal tissues and malignancies in cancer patients and correlate concordance with alphavbeta6 expression.

OUTLINE:

Patients receive 18F-alphavbeta6-BP intravenously (IV) and then undergo positron emission tomography (PET) scans over 30 minutes each at 30, 60, 120, and 180 minutes post-injection.

After completion of study, patients are followed up for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary or metastatic cancer in one or more of the following locations: breast, colorectal, lung, pancreas
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
* Will sign the Institutional Review Board (IRB)-approved consent form
* Able to remain motionless for up to 30-60 minutes per scan

Exclusion Criteria:

* Creatinine > 2 x upper limit of normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2 x upper limit of normal
* Life expectancy < 3 months (mo)
* Women who are pregnant or breast-feeding
* Patients who cannot undergo PET/compute tomography (CT) scanning
* Lack of availability for follow-up assessments
* Participation in another clinical trial involving an investigational agent within 4 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2016-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of safe administration of 18F-αvβ6-BP | Up to 6 months
  Assessed by measures and/or changes in a given vital sign

SECONDARY OUTCOMES:
Measurement of 18F-αvβ6-BP accumulation in tumors | Up to 6 months
  Assessed by PET
Level of αvβ6-BP expression in tumors | Up to 6 months
  Immunohistochemistry (IHC) staining for the cell surface receptor integrin

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sutcliffe, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States